CLINICAL TRIAL: NCT00154882
Title: Weekly Low-dose Paclitaxel (Phyxol) Plus 24-Hour Infusion of Cisplatin as First-line Chemotherapy for Metastatic Breast Cancer
Brief Title: Paclitaxel (Phyxol) and Cisplatin as First-line Chemotherapy for Metastatic Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 920705
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2010-01-21 (Estimated); Status verified 2005-07

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; First-line
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: Paclitaxel (Phyxol) , Cisplatin

INTERVENTIONS:
Drug: Paclitaxel (Phyxol) , Cisplatin

SUMMARY:
The primary endpoint of this phase II trial is the objective response rate of the stage I (low-dose) regimen. The secondary endpoints include treatment-related toxicity, the change in quality of life, progression free survival and overall survival.

DETAILED DESCRIPTION:
Breast cancer is one of the leading causes of cancer death for women in Taiwan. We have recently demonstrated that combination of paclitaxel and cisplatin, at conventional doses, is highly effective in the treatment of breast cancer. However, the acute and cumulative toxicities of paclitaxel have been troublesome to a significant portion of the patients. Several lines of evidence suggested that weekly paclitaxel, at a much lower dose range of 40 to 50 mg/m2 per week, may be as effective as that of the conventional doses of paclitaxel (80 to 90 mg/m2 per week) for patients with metastatic ovarian and lung cancers. The low-dose regimen of paclitaxel may significantly improve the compliance of the patients. This open-label phase II trial is designed to test this hypothesis.

ELIGIBILITY:
Inclusion Criteria:

1. Women with histologically proven breast cancer and clinical evidence of distant metastasis
2. The index lesions should be at least 20 mm × 20 mm in size
3. Age must be older than 18 and younger than 75 year-old
4. Karnofsky performance status > 70%
5. Adequate bone marrow reserves, defined as white blood cell (WBC) > 4,000, absolute neutrophil count (ANC) > 1,500, platelet > 100,000
6. Liver transaminases < 3 times upper normal limit if no liver metastasis and 5 times upper normal limit if liver metastasis is present; total bilirubin < 2 mg/dl; serum creatinine < 1.5 mg/dl
7. No prior chemotherapy for metastatic disease. Previous chemotherapy as adjuvant treatment is acceptable, if the adjuvant chemotherapy has been completed at least 6 months before entry into in this study
8. If the patients have received hormonal therapy for metastatic disease, there must be definite evidence of disease progression under the hormonal therapy, and hormonal therapy should be discontinued before entry into this study
9. Previous or concurrent radiotherapy is acceptable if the area of radiation does not involve the site of the index tumor lesions
10. Patients of childbearing age should have effective contraception during the study period
11. All patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional guidelines.

Exclusion Criteria:

1. Patients who are receiving concurrent hormonal or cytotoxic therapy or other experimental therapy. Concurrent therapy with other biological agents, such as Trastuzumab (Herceptin), is not allowed
2. Patients who refuse port-A catheter implantation
3. Patients who have received taxane (paclitaxel or docetaxel) or cisplatin as adjuvant chemotherapy
4. Patients with brain or leptomeningeal metastases
5. Patients who have significant cardiac arrhythmia or acute myocardial infarction within 6 months before entry
6. Patients who have major systemic diseases that the attending physicians considered inappropriate for systemic chemotherapy
7. Life expectancy less than 2 months
8. Pregnant or nursing patients may not participate. Patients with reproductive potential may not participate unless they have agreed to use an effective contraceptive method
9. No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancers, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any cancer from which the patient has been disease-free for 5 years

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2003-09; Study Completion 2007-07 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint of this phase II trial is the objective response rate of the stage I (low-dose) regimen. | 2003~2008

SECONDARY OUTCOMES:
The secondary endpoints include treatment-related toxicity, the change in quality of life, progression free survival and overall survival. | 2003~2008

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Shen Lu, M.D., Principal Investigator — Department of Oncology , National Taiwan University Hospital
Locations (1):
- Department of Oncology , National Taiwan University Hospital, Taipei, Taiwan